CLINICAL TRIAL: NCT02232360
Title: The Comparative Analysis of the Effects on Plaque Volume and Tissue Characteristics Between Combined Therapy With STAatin Plus FENOfibrate and Statin Alone in Mild to Moderate, Non- Intervened Coronary Artery Stenosis (STAFENO Trial)
Brief Title: Effects of Combined Therapy With Statin Plus Fenofibrate on Coronary Atherosclerotic Plaque Compared With Statin Alone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Seung Hwan Han, Professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAFENO
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
Keywords: Atherosclerotic plaque; Virtual histology intravascular ultrasound; Plaque composition; Rosuvastatin; Fenofibrate; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic | interventions — Rosuvastatin Calcium; Fenofibrate; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin and fenofibrate (Experimental): Combination therapy: rosuvastatin 10 mg and fenofibrate 160 mg per day
  Interventions: Drug: Rosuvastatin and fenofibrate
- Rosuvastatin alone (Active Comparator): Rosuvastatin 10 mg per day
  Interventions: Drug: Rosuvastatin alone

INTERVENTIONS:
Drug: Rosuvastatin and fenofibrate — Combination therapy: rosuvastatin 10 mg and fenofibrate 160 mg per day
  Other Names: Combination therapy with rosuvastatin and fenofibrate
  Arms: Rosuvastatin and fenofibrate
Drug: Rosuvastatin alone — Rosuvastatin 10mg per day
  Other Names: Rosuvastatin alone therapy
  Arms: Rosuvastatin alone

SUMMARY:
The purpose of this study is to determine effects of combination therapy with rosuvastatin and fenofibrate on atheromatous plaques and its tissue characteristics of de novo coronary lesions with intermediate stenosis in patient with coronary artery disease, compared with rosuvastatin alone therapy.

DETAILED DESCRIPTION:
Cardiovascular disease remains the leading cause of morbidity and mortality worldwide. In the past few decades, optimal pharmacological therapies with statins targeting LDL-cholesterol substantially reduce the risks of cardiovascular disease. However, the residual cardiovascular risk is still high, requiring need for additional preventive therapies to achieve even greater risk reduction.

Recent meta-analysis demonstrated fibrates can reduce the risk of coronary events and might have a role in patients with high cardiovascular risks or combined dyslipidemia. Likewise, fenofibrate had a possible benefit for patients with high triglyceride level and low HDL-cholesterol level in the post-hoc analysis of ACCORD or FIELD trials.

Thus, investigators tried to determine effects of combination therapy with rosuvastatin and fenofibrate on atheromatous plaques and its tissue characteristics of de novo coronary lesions with intermediate stenosis in patient with coronary artery disease, compared with rosuvastatin alone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease who were 20 years of age or older and needed coronary angiography
* Intermediate coronary artery stenosis (diameter stenosis ≥30% to ≤60% by visual estimation, diameter ≥2.0 mm to ≤4.0 mm, de novo lesion in native coronary artery) in which virtual histology-intravascular ultrasound (VH-IVUS) could be feasible
* Combined dyslipidemia

  * Stain-naive patients - LDL-cholesterol ≥70 mg/dL and non-HDL-cholesterol ≥130 mg/dL
  * Patients taking statin within 2 weeks - LDL-cholesterol < 100 mg/dL and non-HDL-cholesterol ≥100 mg/dL
* Patients who gave written informed consent

Exclusion Criteria:

* Diabetic patients
* Cardiogenic shock
* Heart failure with symptoms of New York Heart Association class III/IV or left ventricular ejection fraction <35%
* Renal dysfunction (creatinine level ≥1.7 mg/dL or dependence of dialysis
* Hepatic dysfunction (transaminase level > 3 times of normal within limit)
* Pregnancy or breast-feeding women
* Familial hypercholesterolemia
* Hypertriglyceridemia (triglyceride level >500 mg/dL)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percent and Absolute changes of Necrotic Core volume in non-culprit intermediate lesions | After 12±2 months treatment
  Percent and Absolute changes of Necrotic Core volume in non-culprit intermediate lesions by VH-IVUS

SECONDARY OUTCOMES:
Percent and Absolute changes of area of necrotic core, dense calcium, fibrous plaque in non-culprit intermediate lesions | After 12±2 months treatment
  Percent and Absolute changes of area of necrotic core, dense calcium, fibrous plaque in non-culprit intermediate lesions by VH-IVUS
Presence of thin-cap fibroatheroma | After 12±2 months treatment
  change of plaque phenotype by VH-IVUS
Absolute and percent changes of volume/area of external elastic membrane, lumen and plaque volume | After 12±2 months treatment
  Absolute and percent changes of volume/area of external elastic membrane, lumen and plaque volume by VH-IVUS
Remodeling index | After 12±2 months treatment
  Remodeling index by VH-IVUS
Major adverse cardiovascular events (MACE) | After 12 months treatment
  The composites of all-cause death, non-fatal myocardial infarction, stroke, culprit lesion revascularization, or non-culprit lesion revascularization
Adverse drug events | After 12±2 months treatment
  Adverse drug events related by study drugs
Creatine phosphokinase | After 12±2 months treatment
  measurement of muscular side effects related by study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hwan Han, MD, Principal Investigator — Gachon University Gil Medical Center
Locations (6):
- South Korea (6):
  - Konyang University Hospital, Daejeon
  - Chonnam National University Medical School and Hospital, Gwangju
  - Inje University ilsanPaik Hospital, Ilsan
  - Gachon University Gil Medical Center, Incheon
  - Chung-Ang University Hospital, Seoul
  - Seoul National Univesity Boramae Medical Center, Seoul

REFERENCES:
- [Derived] Kwon TG, Jang AY, Kim SW, Hong YJ, Bae JH, Lee SY, Kim SH, Han SH. Design and rationale of a randomized control trial testing the effectiveness of combined therapy with STAtin plus FENOfibrate and statin alone in non-diabetic, combined dyslipidemia patients with non-intervened intermediate coronary artery disease - STAFENO study. Trials. 2020 Apr 22;21(1):353. doi: 10.1186/s13063-020-04291-5. PMID 32321551